CLINICAL TRIAL: NCT03736005
Title: Skeletal Muscle Wasting and Renal Dysfunction in Patients After Critical Illness and Major Trauma - Outcomes Study
Brief Title: Skeletal Muscle Wasting and Renal Dysfunction After Critical Illness Trauma - Outcomes Study
Acronym: KRATOS
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: KRATOSProtocolv1.2
Record Dates: First submitted 2018-08-28; First posted 2018-11-08 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Critical Illness; Acute Kidney Injury; Muscle Loss; Major Trauma; Quality of Life; Chronic Kidney Diseases
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury; Muscular Atrophy; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Quadriceps muscle tissue, blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General ICU admissions: Non- major trauma ICU admission Exposure to significant period of critical illness
  Interventions: Other: Exposure of significant critical illness
- Major Trauma admissions: Exposure to Major Trauma Exposure to significant period of critical illness
  Interventions: Other: Exposure of significant critical illness

INTERVENTIONS:
Other: Exposure of significant critical illness — Exposure. Observational study with all patients invited to follow-up clinic for kidney, muscle and functional assessments.

SUMMARY:
This study aims to determine changes in kidney function during and after critical illness, comparing conventional creatinine based methods with the gold standard to accurately establish the presence of new or worsened chronic kidney disease. In addition, investigators will assess the confounding effect of muscle wasting on the conventional assessment of kidney function and investigate the information that measures of kidney function may contribute to the assessment of musculoskeletal health after critical illness.

DETAILED DESCRIPTION:
More people than ever are surviving life-threatening illnesses such as major trauma. However, until now doctors and researchers have focused more on improving short term survival than on the serious, long-term complications experienced by survivors of critical illness. In response, the National Institute for Health and Care Excellence (NICE) and patient-clinician partnerships such as the James Lind Alliance, have now prioritised research into the diagnosis, follow-up and treatment of critical care survivors.

Development of chronic kidney disease and persistent muscle weakness are two commonly encountered complications which significantly impact long-term health and wellbeing after critical illness. Worsening of kidney function strongly predisposes to development of heart disease, premature death or need for long-term dialysis. Similarly, the muscle wasting experienced by almost all survivors of critical illness can result in persistent, life changing limitations to daily living, inability to work and decreased quality of life. Importantly, the human and economic consequences of critical illness may be particularly profound in major trauma victims who are often young and previously healthy. In this project, investigators will aim to simultaneously measure changes in kidney function and muscle mass after critical illness allowing researchers to understand how these processes interact in affecting longer-term patient outcomes.

The investigators will recruit 62 patients, 31 admitted to intensive care after major trauma and 31 admitted for other reasons. Complementary methods will be used to accurately monitor muscle mass and kidney function. Six months after discharge from hospital, patient's ability to manage their daily activities and quality of life will be assessed alongside measurements of muscle mass, strength and kidney function. The study will be performed at the Royal London Hospital, an internationally renowned centre for critical care and trauma research.

ELIGIBILITY:
Inclusion Criteria:

* Major trauma cohort: Patients ≥18y admitted to ICU and anticipated to be mechanically ventilated for ≥48 hours with a primary admission diagnosis of major trauma.
* Non-trauma cohort: Patients ≥18y admitted to ICU and anticipated to be mechanically ventilated for ≥48 hours without a primary admission diagnosis of major trauma.

Exclusion Criteria:

* Death or discharge from hospital considered highly likely by treating physician within 7 days of ICU admission.
* Any of the following conditions: major traumatic brain injury (Abbreviated Injury Scale head injury score ≥ 5), spinal cord injury with paralysis, lower limb amputation, end stage renal disease or disseminated cancer, lack of independence with activities of daily living or non-ambulatory status prior to admission. (Rationale - exclusion of factors where type of injury or comorbid disease will overwhelming determine functional or renal outcomes.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to critical care.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Change in estimated Glomerular Filtration Rate (eGFR) between creatinine- and cystatin C-based estimates. | At 7 days after ICU discharge.

SECONDARY OUTCOMES:
Rectus Femoris muscle wasting | From ICU admission (day 1 to 10) and 7 days and 6 months after ICU discharge. Time period up to and including 18 months from recruitment.
  Change in cross sectional area of Rectus Femoris assessed via ultrasound
Diagnosis of a negative Nitrogen Balance | From ICU admission (day 1 to 10) and 7 days after ICU discharge.
  Serum and urinary urea measurements aggregated as net nitrogen balance.
Respiratory muscle wasting | From ICU admission (day 1 to 10) and 7 days and 6 months after ICU discharge.
  Change in cross sectional area of intercostal muscle, change in diaphragm thickness
Loss of muscle quality | From ICU admission (day 1 to 10) and 7 days and 6 months after ICU discharge.
  Change in Rectus femoris muscle echogenecity
Loss of functional capacity | 7 days and 6 months after ICU discharge.
  Change in Functional Independence Measure
Diagnosis of Anxiety of Depression | 7 days and 6 months after ICU discharge.
  Change in Hospital Anxiety and Depression Scale
Diagnosis of Sarcopaenia | From ICU admission (day 1 to 10) and 7 days and 6 months after ICU discharge.
  Assessed using bioelectrical impedance analysis, change in cross sectional area of abdominal skeletal muscle,
Diagnosis of Intensive care unit acquired weakness | From ICU admission (day 1 to 10) and 7 days and 6 months after ICU discharge.
  Assessed using MRC Sum score
Diagnosis of Intensive care unit acquired weakness | From ICU admission (day 1 to 10) and 7 days and 6 months after ICU discharge.
  Assessed using hand grip strength.
Change in quality of life | pre-admission baseline then 7 days and 6 months after ICU discharge.
  Change in Euroqol 5d 5L (European quality of life group, quality of life instrument version 5D5L)
Change in walking capacity | 7 days and 6 months after ICU discharge.
  Change in Six minute walk test
Diagnosis of chronic kidney disease | 6 months after ICU discharge
  Diagnosis using creatinine clearance, iohexol and serum creatinine derived eGFR
Diagnosis of non-recovery of eGFR to baseline | From ICU admission (day 3 to 10) and 7 days after ICU discharge.
  Diagnosis using creatinine clearance, iohexol and serum creatinine derived eGFR

CONTACTS AND LOCATIONS:
Locations (1):
- Royal London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ravn B, Prowle JR, Martensson J, Martling CR, Bell M. Superiority of Serum Cystatin C Over Creatinine in Prediction of Long-Term Prognosis at Discharge From ICU. Crit Care Med. 2017 Sep;45(9):e932-e940. doi: 10.1097/CCM.0000000000002537. PMID 28614196
- [Derived] Haines RW, Fowler AJ, Liang K, Pearse RM, Larsson AO, Puthucheary Z, Prowle JR. Comparison of Cystatin C and Creatinine in the Assessment of Measured Kidney Function during Critical Illness. Clin J Am Soc Nephrol. 2023 Aug 1;18(8):997-1005. doi: 10.2215/CJN.0000000000000203. Epub 2023 May 31. PMID 37256861